CLINICAL TRIAL: NCT00543933
Title: Acute Effect of Inhaled Nitric Oxide on Pulmonary Insufficiency in Congenital Heart Disease
Brief Title: Pilot Study of Inhaled Nitric Oxide to Treat Pulmonary Insufficiency in Congenital Heart Disease
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Investigator left institution
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-491
Record Dates: First submitted 2007-10-11; First posted 2007-10-15 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Pulmonary Insufficiency
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Nitric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- iNO administered (Experimental): iNO administered at 40 ppm via a non-rebreather mask
  Interventions: Drug: iNO administered

INTERVENTIONS:
Drug: iNO administered — iNO at 40 ppm through a non-rebreather mask for 5 minutes
  Other Names: Nitric Oxide

SUMMARY:
Inhaled nitric oxide in patients with pulmonic valve insufficiency.

DETAILED DESCRIPTION:
Pulmonic valve insufficiency (PI) is a well-defined problem after primary surgical repair of Tetralogy of Fallot (TOF). Though well-tolerated for years, long-term PI can lead to structural changes in the right ventricle, the sequelae of which include right heart failure, arrhythmia, and sudden cardiac death. The only current treatment for severe symptomatic PI is pulmonic valve replacement. We hypothesize that inhaled nitric oxide (iNO), a selective pulmonary vasodilator, can acutely decrease PI as assessed by cardiac magnetic resonance imaging (CMR). Methods: 22 consecutive patients with PI in the setting of corrected TOF or post pulmonic valve balloon valvuloplasty will undergo a clinically indicated CMR. Nitric oxide gas will be delivered via facemask through a specialized delivery device at 40ppm. After 5 minutes, flow velocity mapping and gradient echo sequences will be repeated to assess pulmonary regurgitant fraction, right ventricular volumes, and ejection fraction. Nitric oxide will be discontinued after acquisition of the last picture. Wilcoxon rank-sum for paired data will be used to assess effect of intervention. Significance: If decreasing pulmonary vascular resistance decreases PI, medical therapy with long-acting pulmonary vasodilators may be an attractive therapeutic option with the goal of delaying or even obviating pulmonic valve replacement.

ELIGIBILITY:
Inclusion Criteria:

* Known pulmonary insufficiency status
* Previous Tetralogy of Fallot repair or balloon valvuloplasty/surgical valvotomy for pulmonary stenosis
* Clinically indicated cardiac magnetic resonance imaging study

Exclusion Criteria:

* Enrollment in another clinical trial
* Age less then 18 years
* Inability to provide informed consent
* Institutionalized individual
* Pregnant or lactating
* Serious claustrophobia
* Pacemaker/ICD
* Aneurysm clips
* Internal hardware
* Severe obesity (>350lbs)
* Residual ventricular septal defect
* History of methemoglobinemia
* History of blood dyscrasias
* Acute pulmonary infection
* Pulmonary edema
* Hypersensitivity to nitric oxide or any of its components
* Left ventricle dysfunction (EF<40%)
* Concurrent use of nitroglycerin or prilocaine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-10 (Actual); Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
pulmonary regurgitant volume and fraction | Single time point
  Aortic regurgitant fraction measured by CMR velocity flow mapping

CONTACTS AND LOCATIONS:
Overall Officials: Richard Krasuski, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hart SA, Devendra GP, Kim YY, Flamm SD, Kalahasti V, Arruda J, Walker E, Boonyasirinant T, Bolen M, Setser R, Krasuski RA. PINOT NOIR: pulmonic insufficiency improvement with nitric oxide inhalational response. J Cardiovasc Magn Reson. 2013 Sep 4;15(1):75. doi: 10.1186/1532-429X-15-75. PMID 24006858